CLINICAL TRIAL: NCT01207284
Title: Influence of Physical Therapy Intervention on the Foot and Ankle in Gait Biomechanics in Individuals With Diabetic Neuropathy: a Randomized Clinical Trial
Brief Title: Influence of Physical Therapy for Foot and Ankle in the Gait of Individuals With Diabetic Neuropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LaBiMPH-001
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Diabetic Neuropathy With Loss of Sensation; Foot and Ankle Muscle Weakness; Foot and Ankle Range of Movement Restriction
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Therapy (Experimental): Foot and ankle passive and active stretching, muscle strengthening, proprioception training and gait training.
  Interventions: Other: Physical Therapy
- Control (No Intervention)

INTERVENTIONS:
Other: Physical Therapy — strengthening passive and active stretching balance training gait training
  Arms: Physical Therapy

SUMMARY:
The hypothesis is that a physical therapy intervention for foot and ankle of diabetic neuropathic individuals would affect positively the way they walk, lowering the harmful forces that these segments receive, that are associated mainly with lower range of movement, muscle weakness and loss of sensation. The participants will be randomly assigned into control group (regular treatment prescribed by their medical group) or into treatment group, that will receive 12 weeks of physical therapy intervention, twice a week, for 45 minutes each session. This will aim for increasing foot and ankle range of movement, muscle strength and improving sensory inputs.

DETAILED DESCRIPTION:
In this study, were included subjects diagnosed with diabetic neuropathy, aged between 45 and 65 years old. We aimed to assess the effect of a physical therapy program on biomechanics of lower limbs during gait.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 1 or 2 diagnosed for at least seven years
* body mass index ranging 18.5-29.9 kg/m2 (normal and overweight classifications)
* diabetic polyneuropathy diagnosed by the medical care center: score higher than 2 out of 13 in the Michigan Neuropathy Screening Instrument (MNSI) questionnaire, indicating the presence of at least two diabetic polyneuropathy symptoms; score higher than 1 out of 10 for physical assessment of the MNSI instrument, but always including impaired vibration perception
* ability to walk independently in the laboratory

Exclusion Criteria:

* ulceration not healed for at least 6 months
* partial or total foot amputation
* receiving any physiotherapy intervention or offloading devices
* neurological or orthopedic impairments
* major vascular complications
* severe retinopathy
* severe nephropathy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Peak pressure at lateral forefoot | 12 weeks

SECONDARY OUTCOMES:
Peak pressure | 12 weeks
  In 5 foot areas: heel, midfoot, medial forefoot, hallux and toes.
Peak pressure | 24 weeks
  In foot areas: heel, midfoot, medial forefoot, lateral forefoot, hallux and toes.
Time-to-peak pressure | 12 weeks
  In 6 foot areas: heel, midfoot, lateral forefoot, medial forefoot, hallux and toes.
Time-to-peak pressure | 24 weeks
  In 6 foot areas: heel, midfoot, lateral forefoot, medial forefoot, hallux and toes.
Pressure-time integral | 12 weeks
  In 6 foot areas: heel, midfoot, lateral forefoot, medial forefoot, hallux and toes.
Pressure-time integral | 24 weeks
  In 6 foot areas: heel, midfoot, lateral forefoot, medial forefoot, hallux and toes.
Mean velocity of center of pressure displacement | 12 weeks
  In 7 foot areas: heel, midfoot, lateral forefoot, medial forefoot, hallux, toes and total area.
Mean velocity of center or pressure displacement | 24 weeks
  In 7 foot areas: heel, midfoot, lateral forefoot, medial forefoot, hallux, toes and total area.
Sagittal range of motion of ankle | 12 weeks
Sagittal range of motion of ankle | 24 weeks
Sagittal peak of extensor moment of ankle | 12 weeks
Sagittal peak of extensor moment of ankle | 24 weeks
Sagittal peak of flexor moment of ankle | 12 weeks
Sagittal peak of flexor moment of ankle | 24 weeks
Michigan Neuropathy Screening Instrument score for symptoms | 12 weeks
Michigan Neuropathy Screening Instrument score for symptoms | 24 weeks
Michigan Neuropathy Screening Instrument score for physical assessment | 12 weeks
Michigan Neuropathy Screening Instrument score for physical assessment | 24 weeks
Functional tests score | 12 weeks
Functional tests score | 24 weeks
Muscle function score | 12 weeks
Muscle function score | 24 weeks
Activities-Specific Balance Confidence Scale (ABC) | 12 weeks
Activities-Specific Balance Confidence Scale (ABC) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Isabel CN Sacco, Study Chair — University of Sao Paulo
Locations (1):
- Department of Speech, Physical Therapy and Occupational Therapy, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sartor CD, Hasue RH, Cacciari LP, Butugan MK, Watari R, Passaro AC, Giacomozzi C, Sacco IC. Effects of strengthening, stretching and functional training on foot function in patients with diabetic neuropathy: results of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 27;15:137. doi: 10.1186/1471-2474-15-137. PMID 24767584
- [Derived] Sartor CD, Watari R, Passaro AC, Picon AP, Hasue RH, Sacco IC. Effects of a combined strengthening, stretching and functional training program versus usual-care on gait biomechanics and foot function for diabetic neuropathy: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Mar 19;13:36. doi: 10.1186/1471-2474-13-36. PMID 22429765